CLINICAL TRIAL: NCT03275753
Title: Visual Function Tests in Non-Exudative Age-Related Macular Degeneration and Normal Subjects
Brief Title: Visual Function Tests in Age-related Macular Degeneration
Status: Terminated | Type: Observational
Why Stopped: Study terminated by Sponsor
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-270-0001
Record Dates: First submitted 2017-08-08; First posted 2017-09-08 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Age Related Macular Degeneration
Keywords: Visual function; Critical flicker fusion; Dark adaptation; Reading test
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal Population: VA of 20/25 or better in the study eye with no prior diagnosis of any retinal or ocular diseases
  Interventions: Other: Visual Function Tests
- Early Dry AMD Population: VA of 20/40 or better in the study eye with clinical diagnosis of early dry AMD
  Interventions: Other: Visual Function Tests
- Intermediate Dry AMD Population: VA of 20/40 or better in the study eye with clinical diagnosis of intermediate dry AMD
  Interventions: Other: Visual Function Tests
- Advanced Dry AMD Population: Clinical diagnosis of advanced dry AMD in the study eye
  Interventions: Other: Visual Function Tests

INTERVENTIONS:
Other: Visual Function Tests — All subjects will undergo a battery of visual function tests

SUMMARY:
The goal of this study is to assess a battery of visual function tests in subjects with non-exudative age-related macular degeneration

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is one of the leading causes of visual impairment among elderly populations in developed countries. Majority of AMD patients (80%) suffer from the dry or non-exudative form of the disease. Currently there are no approved treatments for dry AMD. Clinical development of therapeutic agents for dry AMD is limited by slow progressing nature of the disease as well as the lack of sensitive endpoints to assess therapeutic efficacy. Visual acuity, the commonly used functional endpoint, remains minimally affected during early stages of dry AMD. Thus novel visual function endpoints, that can identify functional deficits during early stages of dry AMD prior to development of geographic atrophy, are needed. In the current study a battery of visual function tests will be evaluated in subjects with different stages of dry AMD and normal controls, to assess their sensitivity and feasibility as potential functional endpoints for dry AMD.

ELIGIBILITY:
Inclusion Criteria:

* All Subjects Must:

  1. Be 60 years of age or older;
  2. Provide written informed consent;
  3. Be willing and able to follow all instructions and attend the study visits;
  4. Must be able to perform all study procedures;

     Normal Subjects:
  5. Have BCVA of 20/25 or better in the study eye;
  6. Have no history or clinical evidence of AMD, retinal diseases or any other ocular pathologies in either eye;

     AMD Subjects:
  7. Have BCVA of 20/40 or better in the study eye;
  8. Have a clinical diagnosis of non-exudative AMD in the study eye;

     Exclusion Criteria:

     All subjects must not have any of the below criteria

  <!-- -->

  1. Have a diagnosis of wet AMD in the study eye;
  2. Have any other hereditary or acquired retinal diseases in either eye ;
  3. Have glaucoma or other optic nerve diseases in either eye;
  4. Have corneal or other anterior segment diseases in either eye;
  5. Have significant cataract in the study eye;
  6. Have a history of ocular trauma or ocular surgery (other than cataract removal) in the study eye;
  7. Have a history of uncontrolled systemic disease (e.g. poorly controlled hypertension or poorly controlled diabetes);
  8. Have a history of seizures;
  9. On psychotropic medications;
  10. Any other symptoms or conditions that could, in the opinion of the investigator, interfere with study procedures.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Normal Population (N=50) VA of 20/25 or better in the study eye with no prior diagnosis of any retinal or ocular diseases.
  Group 2: Early Dry AMD Population (N=50) VA of 20/40 or better in the study eye with clinical diagnosis of early dry AMD based on fundus features.
  Group 3: Intermediate Dry AMD Population (N=50) VA of 20/40 or better in the study eye with clinical diagnosis of intermediate dry AMD based on fundus features.
  Group 4: Advanced Dry AMD Population (N=50) Clinical diagnosis of advanced dry AMD based on fundus features in the study eye
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Critical flicker fusion | At study visit through study completion, an average of 2 years
  Critical flicker fusion will be tested using a computer based test for different stimulus colors, white, red, green and blue. A wide range of luminance and contrast levels will be tested. The subject would be seated in front of the monitor. The non-study eye will be occluded. Subjects would be given adequate practice tests prior to performing the actual test. The stimulus will be presented on the monitor screen and the subject indicates perceiving the stimulus by pressing a test button.

SECONDARY OUTCOMES:
Dark adaptation | At study visit through study completion, an average of 2 years
  Dark adaptation function will be assessed with dilated pupils using computer based stimuli following photo bleach. Subject will be seated in front of the test monitor with best correction in place for the study eye. The subject will be instructed to keep fixating on a red fixation cross in the center of the monitor and respond to perceiving the stimulus presented by pressing the response trigger button. All stimuli will be presented in random order for all intensities presented. The stimulus intensity is programmed to decrease in intensity with time. The test will be terminated after 20 minutes of recording. Dark adaptation curve will be generated and rod-cone recovery time (in minutes) will be derived from the curve.
Reading Tests | At study visit through study completion, an average of 2 years
  Reading tests will be performed using an electronic tablet device. The subject will be seated in a comfortable position with the non-tested eye occluded. The tablet will be set up in a table right in front of the subject at a viewing distance of 40cm. The subject will be given detailed instructions on the test procedures and outcomes. The goal of this test to assess reading speed of the study eye under a variety of conditions such as high contrast-high luminance, low contrast, low luminance, crowded letters, pepper words of different lengths and vanishing optotypes. Each challenge will be tested using a different passage of similar difficulty level. For each passage, reading speed will be estimated as the time taken to accurately read the entire passage and recorded in words per minute (WPM).
Color vision function | At study visit through study completion, an average of 2 years
  Color vision function will be assessed to test L, M and S cone functions. During the test, a letter will briefly flash on the screen. The subject then must verbally identify the letter and/or its orientation. The response of the subject is then recorded by the technician. If correct, the next letter is presented at decreased color contrast relative to the background. The test continues in this manner until the subject incorrectly identifies the presented letter. At that point, the stimulus is presented at the next higher contrast level. This continues until the subject correctly identifies the presented letter. The test then terminates.
Shape discrimination | At study visit through study completion, an average of 2 years
  Shape discrimination will be tested by presenting a two-alternative forced choice stimulus to the subject on a computer device (monitor or tablet). The subject will be asked to identify the stimulus which is modulated and which is not. The test shall be performed at full room lighting for photopic sensitivity as well as in reduced lighting (mesopic) conditions. The effect of eccentricity may be tested by presenting successively larger targets with foveal fixation.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chin, OD, Principal Investigator — ORA, Inc.
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No